CLINICAL TRIAL: NCT05977088
Title: Prediction of Cognitive, Neurotrophic, Anti-Inflammatory, and Antioxidant Effectiveness of rTMS Application in Alzheimer's Patients
Brief Title: Prediction of Effectiveness of rTMS Application in Alzheimer's Patients
Acronym: PRIM-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Bezmialem Vakif University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Prof Dr MD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 221S749
Record Dates: First submitted 2023-06-02; First posted 2023-08-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; TMS-EEG; Anti-inflammatory-neuroprotective-antioxidant effect
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): Power Mag TMS device will be used throughout the study, and the excitations will be made with the help of an 8 shaped coil (diameter: 70 mm) with internal cooling. The right-left DLPFC, which is the application area, will be determined with the help of the primary motor hand area and the 10/20 EEG system.
  A resting state EEG (eyes open-closed) will be taken i in the Faraday cage.
  Interventions: Device: Repetetive Transcranial Magnetic Stimulation
- Sham (Sham Comparator): The same treatment procedures will be applied to the control group with a sham coil.
  Interventions: Device: Repetetive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetetive Transcranial Magnetic Stimulation — .Power Mag TMS device will be used throughout the study, and the excitations will be made with the help of an 8 shaped coil (diameter: 70 mm) with internal cooling. The right-left DLPFC, which is the application area, will be determined with the help of the primary motor hand area and the 10/20 EEG system.
  A resting state EEG (eyes open-closed) will be taken in the Faraday cage. The same procedures will be done with the sham coil in the control group.
  Other Names: Electroensefolography

SUMMARY:
Since pharmacological methods are insufficient in the treatment processes of Alzheimer's disease, non-pharmacological methods such as Transcranial Magnetic Stimulation (TMS) have started to be tried as a treatment option as in other neurological and psychiatric diseases. Repeated (rTMS) offers a potential treatment pathway for neurological and psychiatric illnesses. rTMS benefit rate may vary depending on many factors such as the region where it is applied, the progression and the disease degree. The possible effects of TMS on Alzheimer's pathophysiology and modification of disease process (neuroprotective, anti-inflammatory and antioxidant) will also be revealed through blood samples taken from patients before and after treatment. These approaches also constitute the original value of our study.

DETAILED DESCRIPTION:
Since pharmacological methods are insufficient in the treatment processes of Alzheimer's disease, non-pharmacological methods such as Transcranial Magnetic Stimulation (TMS) have started to be tried as a treatment option as in other neurological and psychiatric diseases. Repeated (rTMS) offers a potential treatment pathway for neurological and psychiatric illnesses. rTMS benefit rate may vary depending on many factors such as the region where it is applied, the progression and the disease degree. This study aim is to predict the benefit rate to be obtained from the treatment by using various evaluation parameters before starting rTMS treatment. The possible effects of TMS on Alzheimer's pathophysiology and modification of disease process (neuroprotective, anti-inflammatory and antioxidant) will also be revealed through blood samples taken from patients before and after treatment. These approaches also constitute the original value of our study.

In our project, 20 people will be included in the study and control groups and electroencephalography (EEG) and TMS will be used together in the study. Before rTMS treatment, resting EEG data will be taken for 5 minutes, eyes open and closed. At the end of all these procedures, rTMS treatment will be started, which will take 5 days. The treatment will consist of two sessions per day with a 20 Hz stimulating protocol, 1500 beats to right-left DLPFC, and totaly 3000 beats. EEG recordings will be taken again from all patients one week after the treatment.

Changes in the cognitive functions of Alzheimer's patients will be made through the neuropsychometric test battery taken before and after rTMS. With the analysis of neuropsychometric data, the study group will be divided into two subgroups that benefit from TMS and those who do not. In addition, EEG data obtained before and after-TMS will be compared with power spectrum, coherence, functional connectivity and graph methods in both the study and control groups, and information about the electrophysiological effects of TMS will be obtained.

Blood samples of the patients before and after rTMS will be taken and the changes in the metabolites given below will be compared: Brain Derived Neurotrophic Factor, Glial Based Neurotrophic Factor, Total Oxidant Level, Total Antioxidant Level, Oxidative Stress Index, Total Thiol, Native Thiol, Disulfide, Exosome, Inflammation Biomarkers (interleukin 1 Beta, interleukin 6, Tumor Necrosis Alpha, Interferon gamma, Nuclear factor kappa ß), Albumin Globulin ratio, Omega 6 and Omega 3. Thus, rTMS has possible neuroprotective, anti-inflammatory and antioxidant effects, consequently modifying the disease process. Additional information will be obtained about.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with clinical Alzheimer's Disease in accordance with the NINCDS-ADRDA diagnostic criteria
* >55 years old
* Clinical Dementia Rating Scale (CDR) score in the 1-2 range
* Not having any other disease that affects their cognitive functions
* Volunteer to participate in the study

Exclusion Criteria:

* Participant or relative does not give consent
* The patient's inability to participate in the entire study procedure (eg living in another city)
* The patient's history of head trauma with alcohol/substance abuse
* Presence of severe stroke and other neurological sequelae disease in the participant
* Presence of a metal implant on the head or having a pacemaker and contraindications for other TMS applications During the study or 1 month before, having/been receiving/receiving an investigational drug targeting Alzheimer's disease or neuromodulation treatment such as tDCS and TMS, other than standard treatment for AD symptom control such as acetylcholine esterase and memantine, with the potential to affect the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Mini Mental State Examination | Changes Before Treatment and 1 month after treatment
  Cognitive Neuropsychological Test Score
Neuropsychiatric Inventory | Changes Before Treatment and 1 month after treatment
  Cognitive Neuropsychological Test Score
Alzheimer's Disease Assessment Scale | Changes Before Treatment and 1 month after treatment
  Cognitive Neuropsychological Test Score
ADSL | Changes Before Treatment and 1 month after treatment
  Cognitive Neuropsychological Test Score
Geriatric Depression Scale | Changes Before Treatment and 1 month after treatment
  Cognitive Neuropsychological Test Score

SECONDARY OUTCOMES:
Blood samples ELISA analyses | Changes Before Treatment and 1 month after treatment
  BDNF:measured spectrophotometrically with commercially purchased ELISA kits. GDNF:measured spectrophotometrically with commercially purchased ELISA kits. Exosome: measured spectrophotometrically with commercially available ELISA kits.
  Anti-inflammatory Cytokines: IL-1β, IL-6, TNF-α, IFNy, NF-kβ values will be measured spectrophotometrically with commercially purchased ELISA kits.
Blood samples analyses | Changes Before Treatment and 1 month after treatment
  OSI:TOS and TAS will be measured by photometric methods. OSI will be found by mathematical calculation. Total thiol and native thiol concentrations are measured spectrophotometrically in separate solutions prepared for the determination of the thiol-disulfite ratio, which is another indicator of oxidative stress, and the amount of disulfide is determined according to the mathematical ratio between them.
  Albumin Globulin Ratio:measured by electrophoresis method and albumin globulin ratio will be determined.
  Omega 6/3 Levels:determined by commercially purchased lipid mediators.
Inflammatory Biomarker analyses | Changes Before Treatment and 1 month after treatment
  Inflammatory parameters IL-1β, IL-6 and TNF-α will be measured IL-1β, IL-6 and TNF-α levels will be measured photometrically with commercially available ELISA kits.
Oxidative Stress Biomarker analyses | Changes Before Treatment and 1 month after treatment
  TAS, TOS, TT and NT levels of oxidative stress parameters in blood samples taken from AD patients will be measured. TAS, TOS, TT, NT levels of blood samples taken will be measured by photometric method with kits to be purchased commercially. The oxidative stress index (OSI) will be found as TOS/TAS, and the amount of dynamic disulfide bonds will be found by determining half of the difference between the TT and NT groups.
Evaluation of Fatty Acid Profile Analysis with GC-MS | Changes Before Treatment and 1 month after treatment
  Fatty acids comprising more than 95% of the fatty acids detectable in plasma will be measured.
  Tetradecanoic acid,9(Z)-Tetradecenoic acid,Hexadecanoic acid,9(Z)-Hexadecenoic acid,9(E)-Hexadecenoic acid,Octadecanoic acid,9(Z)-Octadecenoic acid,Methyl 9(E)- Octadecenoate,11(Z)-Octadecenoic acid,Methyl 11(E)- Octadecenoate,Methyl 6(Z)- Octadecenoate,9(Z),12(Z)- Octadecadienoic acid,9(E),12(E)- Octadecadienoic acid,9(Z),12(Z),15(Z)- Octadecatrienoic acid, 6(Z),9(Z),12(Z)- Octadecatrienoic acid,Eicosanoic acid,8(Z),11(Z),14(Z)- Eicosatrienoic acid, 5(Z),8(Z),11(Z),14(Z)-Eicosatetraenoic acid, 11(Z)-Eicosenoic acid, 11(Z),14(Z)- Eicosadienoic acid, 5(Z),8(Z),11(Z),14(Z),17(Z)- Eicosapentaenoic acid, Docosanoic acid, 13(Z)-Docosenoic acid 4(Z),7(Z),10(Z),13(Z),16(Z),19(Z)- Docosahexaenoic acid 7(Z),10(Z),13(Z),16(Z)-Docosatetraenoic acid 7(Z),10(Z),13(Z),16(Z),19(Z)- Docosapentaenoic acid 4(Z),7(Z),10(Z),13(Z),16(Z)- Docosapentaenoic acid Tetracosanoic acid 15(Z)-Tetracosenoic acid
Metabolomics Analysis by Liquid Chromatography-Mass Spectrometer/Mass Spectrometer (LC-MS/MS) | Changes Before Treatment and 1 month after treatment
  The 41 amino acids to look for by LC-MS/MS are:
  1. 1-Methylhistidine
  2. 2-Aminoadipic Acid
  3. 3-Aminoisobutyric Acid
  4. 3-Methylhistidine
  5. 4-Hydroxyproline
  6. 5-Hydroxylysine
  7. Alanine
  8. Alloisoleucine
  9. Anserine
  10. Arginine
  11. Argininosuccinic Acid
  12. Asparagine
  13. β-Alanine
  14. Carnosine
  15. Citrulline
  16. Cystine
  17. Cystathionine
  18. Ethanolamine
  19. Gamma-Aminobutyric Acid
  20. Glutamine
  21. Glutamic Acid
  22. Histidine
  23. Homocitrulline
  24. Isoleucine
  25. Leucine
  26. Lysine
  27. Methionine
  28. Norvaline
  29. O-Phosphorylethanolamine
  30. O-Phosphoserine
  31. Ornithine
  32. Phenylanalanine
  33. Proline
  34. Sarcosine
  35. Serine
  36. Taurine
  37. Threonine
  38. Trans-4-Hydroxyproline
  39. Tryptophan
  40. Tyrosine
  41. Valine
EEG Power Spectrum Analysis | Changes Before Treatment and 1 month after treatment
  EEG data will be separated into one-second epochs after they are cleared of noise. Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform (FFT, Fast Fourier Transform) with 10% Hanning window, then power spectrum analysis will be performed, giving the frequency values for each electrode by averaging all FFTs. Maximum peaks will be determined in the delta (0.5-3.5 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (15-28 Hz) and gamma (28-48 Hz) frequency bands. these values will be used in statistical analysis for each person and electrode.
EEG Coherence Analysis | Changes Before Treatment and 1 month after treatment
  Coherence measurements at delta, theta, alpha, beta and gamma frequencies can be analyzed for either intra-hemispheric electrode connections or inter-hemipheric electrode connections.Coherence values take values between 0-1. Values close to 0 indicate that there is no connection at the determined frequency between the two calculated electrode regions, while values close to 1 indicate a high coupling between the two electrode regions. Coherence values will be calculated with the Brain Vision Analyzer program using the formula below.The data obtained during memory and visualization will be separated into one-second epochs after they are cleared of noise.Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform with 10% Hanning window.Then, these data will be calculated for all possible electrode pairs using the brain vision analysis program with the formula given below.

CONTACTS AND LOCATIONS:
Overall Officials: Lutfu Hanoglu, Prof. DR. MD, Principal Investigator — Medipol University
Locations (1):
- Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to ethical reasons